CLINICAL TRIAL: NCT00920426
Title: A Phase 2a Study to Compare Antiviral Effect, Safety, Tolerability and Pharmacokinetics of GSK1265744 Monotherapy Versus Placebo in HIV-1 Infected Adults (ITZ112929)
Brief Title: Study to Compare the Safety and Anti-HIV Effect of GSK1265744 Versus Placebo in HIV-1 Infected Adults (ITZ112929)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112929
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: HIV; naive; Phase II; integrase inhibitor; GSK1265744; newly diagnosed; pharmacokinetics; AIDS; integrase; HIV Infections; Treatment naive
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK1265744 30 mg (Experimental): GSK1265744 30 mg
  Interventions: Drug: GSK1265744 30mg
- Placebo (Experimental): Placebo to match GSK1265744
  Interventions: Drug: Placebo
- GSK1265744 5 mg (Experimental): GSK1265744 5 mg
  Interventions: Drug: GSK1265744 5mg

INTERVENTIONS:
Drug: GSK1265744 30mg — GSK1265744 30 mg
  Arms: GSK1265744 30 mg
Drug: Placebo — Placebo to match GSK1265744
  Arms: Placebo
Drug: GSK1265744 5mg — GSK1265744 5mg
  Arms: GSK1265744 5 mg

SUMMARY:
The purpose of this randomized, double-blinded study is to test the safety of GSK1265744 and how well it works on reducing the amount of HIV in the blood. It will also look at how people react to and how a human body uses GSK1265744. This study will compare the effects of GSK1265744 and placebo.

The study will consist of 1 or 2 parts to look at doses of GSK1265744. About 8 people will take part in Part 1 of the study receiving dose A. If additional dosing information is needed after Part 1, about 6 people will take part in Part 2 of the study receiving dose B.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential, defined as:
* Pre-menopausal females with a documented bilateral oophorectomy, tubal ligation or hysterectomy; or
* Postmenopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone level will be performed to confirm post-menopausal status. For this study, FSH levels > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* CD4+ cell count greater than or equal to 200 cells/mm3 and plasma HIV-1 RNA greater than or equal to 5000 copies/mL at Screening.
* No current antiretroviral therapy and have not received any in the 12 weeks prior to first dose.
* For subjects who have received antiretroviral treatment in the past, adequate treatment options to construct HAART therapy with at least 3 active antiretrovirals for Optimized Therapy, as selected by the Investigator.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* A positive screening Hepatitis B surface antigen; positive screening hepatitis C virus (HCV) antibody and detectable HCV ribonucleic acid (RNA) on subsequent testing. If the hepatitis C antibody is positive but the HCV RNA is undetectable, the subject may be included in the study.
* AST and ALT > 3ULN at Screening. A single repeat is allowed for eligibility determination.
* Inadequate renal function at Screening, defined as either a serum creatinine >1.5 mg/dL or a calculated creatinine clearance (CrCl) ≤ 50 mL/min. A single repeat serum creatinine is allowed to determine eligibility.
* Any acute laboratory abnormality at screening which, in the opinion of the investigator, should preclude the subject's participation in the study of an investigational compound. Any grade 4 laboratory abnormality at screening, with the exception of CPK, will exclude a subject from study participation unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat is allowed for eligibility determination.
* A positive drug screen at screening and baseline. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine or PCP.
* History of regular alcohol consumption, defined as an average weekly intake of >14 drinks for males or >7 drinks for females, within 6 months of Screening.

Note: One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.

* Any condition (including alcohol or drug abuse) which, in the opinion of the investigator, could interfere with the subject's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the subject.
* Prior treatment with an integrase inhibitor (greater than or equal to 1 dose).
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 30 days of study drug administration or anticipated need for such treatment within the study.
* Treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (such as hydroxyurea or foscarnet) within 30 days of study drug administration.
* Treatment with any vaccine within 30 days prior to receiving study medication.
* An active Center for Disease Control and Prevention (CDC) Category C disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Use of multivitamins or antacids within 24 hours prior to the first dose of investigational product.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.

Note: Study medications refer to GSK1265744 or placebo.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* History of clinically relevant pancreatitis or hepatitis within the previous 6 months.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs.
* Exclusion Criteria for Screening ECG (A single repeat is allowed for eligibility determination):

Exclusion Criteria for Screening ECG:

Males Females Heart rate <45 and >100 bpm <50 and >100 bpm QRS duration >120 msec >120 msec QTc interval (Bazett) > 450 msec > 450 msec Non-sustained (≥ 3 consecutive beats) or sustained ventricular tachycardia. Sinus Pauses >3 seconds. 2nd degree (Type II) or higher AV block. Evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes (except early repolarization)).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06-09 (Actual); Primary Completion 2009-08-13 (Actual); Study Completion 2009-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (4):
- United States (4):
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Charlotte, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 centers in the United States from 09 June 2009 to 13 August 2009.
Pre-assignment Details: A total of 9 participants were randomized in the current study to receive 5 milligrams (mg) of GSK1265744 or Placebo. A total of 8 participants were previously randomized in study ITZ111451 part C HIV cohort, NCT00659191 to receive 30 mg of GSK1265744 once daily.
Groups:
- GSK1265744 30 mg: GSK1265744 30 mg once daily was previously studied in study ITZ111451 part C HIV cohort, NCT00659191. Eligible participants received repeat doses of GSK1265744 30 mg (6x5 mg) oral tablets once daily for 10 days.
- GSK1265744 5 mg: Eligible participants received double-blind GSK1265744 5 mg oral tablet once daily for 10 days.
- Placebo: Eligible participants received double-blind matching Placebo oral tablet once daily for 10 days.
- Optimized Therapy: Participants were given investigator chosen optimized therapy for 14 days after being dosed with the randomized regimen (either 5 mg GSK1265744 or Placebo) for 10 days. Participants were unblinded on Day 11 so that the participants receiving Placebo could decline optimized therapy.
Period: ITZ111451
Arm/Group | GSK1265744 30 mg | GSK1265744 5 mg | Placebo | Optimized Therapy
Started | 8 | 0 | 0 | 0
Completed | 7 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: ITZ112929: Randomized Regimen
Arm/Group | GSK1265744 30 mg | GSK1265744 5 mg | Placebo | Optimized Therapy
Started | 0 | 7 | 2 | 0
Completed | 0 | 7 | 2 | 0
Not Completed | 0 | 0 | 0 | 0
Period: ITZ112929: Optimized Therapy (OT)
Arm/Group | GSK1265744 30 mg | GSK1265744 5 mg | Placebo | Optimized Therapy
Started | 0 | 0 | 0 | 8 (Out of 9 participants receiving randomized regimen, 8 participants continued to receive OT.)
Completed | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1265744 30 mg | GSK1265744 5 mg | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 2 | 17
Age, Customized [Count of Participants; unit: Participants]
  27 to 51 Years | 8 | 7 | 2 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 2
  Male | 8 | 5 | 2 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 8 | 5 | 2 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Human Immunodeficiency Virus (HIV-1) Ribonucleic Acid (RNA) to Day 11
Description: Plasma for quantitative HIV-1 RNA was collected on Day 1, 2, 3, 4, 7, 8, 9, 10 and 11. On Days 1, 10 and 11, two samples for HIV-1 RNA was collected between 5-20 minutes apart to reduce sample variability. An HIV-1 RNA PCR assay with a lower limit of detection (LLOD) of 50 copies/milliliter (mL) (ultrasensitive assay) was used for post-baseline assessments. An HIV-1 RNA PCR assay with a LLOD of 400 copies/mL (standard assay) was used for screening and Baseline assessments and included a re-test with and ultrasensitive assay for all Baseline values below the LLOD. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 11
Population: Intent-to-treat (ITT) population comprised of all participants who met study criteria and randomized into study with documented evidence of having received at least 1 dose of randomized treatment and at least 1 post-baseline HIV-1 RNA measurement. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
log10 copies/mL | -2.169 (0.2405) | -0.092 (0.1499)
Statistical Analysis 1: Comparison: GSK1265744 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Analysis of covariance (ANCOVA) with treatment as fixed effect, and Baseline HIV-1 RNA as covariate; Mean Difference (Net) = -2.090, 95% CI 2-sided [-2.547 to -1.632]

2. Primary Outcome: GSK1265744 Pharmacokinetic (PK) Parameters Following Dose Administration on Day 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Within a Participant Across All Treatments(AUC[0-24])
Description: Blood samples for PK analysis of AUC(0-24) of GSK1265744 was collected on Day 1 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose). Samples were collected at nominal times relative to the proposed time of GSK1265744 dosing. The actual date and time of each blood sample collection was recorded. AUC was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: Day 1 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose)
Population: PK Summary Population included participants with evaluable PK profile of GSK1265744 on Day 10. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter (hr*µg/mL)
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 7
Hour*microgram per milliliter (hr*µg/mL) | 7.53 (23)

3. Primary Outcome: GSK1265744 PK Parameters Following Dose Administration on Day 1: Concentration at 24 Hours Post Dose (C24)
Description: Blood samples for PK analysis of C24 of GSK1265744 was collected on Day 1 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose). Samples were collected at nominal times relative to the proposed time of GSK1265744 dosing. The actual date and time of each blood sample collection was recorded.
Time Frame: Day 1 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose)
Population: PK summary population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (µg/mL)
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 7
Micrograms per milliliter (µg/mL) | 0.23 (28)

4. Primary Outcome: GSK1265744 PK Parameters Following Dose Administration on Day 10: Area Under the Concentration-time Curve Over the Dosing Interval (AUC[0-tau])
Description: Blood samples for PK analysis of C24 of GSK1265744 was collected on Day 10 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose). Samples were collected at nominal times relative to the proposed time of GSK1265744 dosing. The actual date and time of each blood sample collection was recorded. AUC was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: Day 10 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µg/mL
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 7
hr*µg/mL | 17.74 (31)

5. Primary Outcome: GSK1265744 PK Parameters Following Dose Administration on Day 10: Predose Concentration (C0), Concentration at End of Dosing Interval (Ctau), Minimum Observed Concentration During One Dosing Interval (Cmin)
Description: Blood samples for PK analysis of C0, Ctau and Cmin of GSK1265744 was collected on Day 10 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose). Samples were collected at nominal times relative to the proposed time of GSK1265744 dosing. The actual date and time of each blood sample collection was recorded.
Time Frame: Day 10 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 7
µg/mL
  C0 | 0.54 (36)
  Ctau | 0.57 (33)
  Cmin | 0.53 (35)

6. Primary Outcome: GSK1265744 PK Parameters Following Dose Administration on Day 1 and Day 10: Maximum Observed Concentration (Cmax)
Description: Blood samples for PK analysis of Cmax of GSK1265744 was collected at pre-dose (within 15 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose on Days 1 and 10. Samples were collected at nominal times relative to the proposed time of GSK1265744 dosing. The actual date and time of each blood sample collection was recorded.
Time Frame: Pre-dose (within 15 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose on Days 1 and 10
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 7
µg/mL
  Day 1 | 0.52 (20)
  Day 10 | 1.02 (25)

7. Primary Outcome: GSK1265744 PK Parameters Following Dose Administration on Day 1 and Day 10: Time to Cmax (Tmax)
Description: Blood samples for PK analysis of tmax of GSK1265744 was collected at pre-dose (within 15 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose on Days 1 and 10. Samples were collected at nominal times relative to the proposed time of GSK1265744 dosing. The actual date and time of each blood sample collection was recorded.
Time Frame: Pre-dose (within 15 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose on Days 1 and 10
Population: as for outcome 3
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 7
Hour
  Day 1 | 2.00 [1.00 to 4.08]
  Day 10 | 2.00 [1.50 to 4.08]

8. Primary Outcome: GSK1265744 PK Parameters Following Dose Administration on Day 1 and Day 10: Terminal Half-life (t1/2) and Absorption Lag Time (Tlag)
Description: PK sampling was planned to be collected up to 24 hours only on Day 1 and Day 10. The data for this outcome measure was however not collected.
Time Frame: Day 1 and Day 10
Population: PK Summary Population. Data for this outcome measure was not collected. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 0

9. Primary Outcome: GSK1265744 PK Parameters Following Last Repeat Administration on Day 10: Apparent Clearance Following Oral Dosing (CL/F)
Description: Blood samples for PK analysis of CL/F of GSK1265744 was collected on Day 10 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose). Samples were collected at nominal times relative to the proposed time of GSK1265744 dosing. The actual date and time of each blood sample collection was recorded.
Time Frame: Day 10 (Pre-dose [within 15 minutes prior to dosing] and at 0.5, 1, 1.5, 2, 3, 4, 6, and 8hours post-dose)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 7
Liter per hour (L/hr) | 0.28 (31)

10. Primary Outcome: Number of Participants With Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, medically significant or is associated with liver injury and impaired liver function.
Time Frame: Day 1 to Day 11
Population: Safety population was defined as all participants who were randomized into the study with documented evidence of having received at least 1 dose of randomized treatment. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 5 mg | Placebo | Optimized Therapy
Number analyzed (Participants) | 7 | 2 | 8
Participants
  Any AEs | 0 | 2 | 3
  Any SAEs | 0 | 0 | 0

11. Primary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils (ANC- Absolute Neutrophil Count), White Blood Cell Count
Description: Blood samples for assessment of hematology parameters of basophils, eosinophils, lymphocytes, monocytes, total neutrophils (ANC- absolute neutrophil count) and white blood cell count was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: Safety population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Thousand cells per microliter
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Thousand cells per microliter
  Basophils, Day 3 | 0.017 (0.0287) | 0.005 (0.0071)
  Basophils, Day 7 | 0.007 (0.0125) | 0.015 (0.0071)
  Basophils, Day 10 | 0.009 (0.0146) | 0.020 (0.0000)
  Eosinophils, Day 3 | -0.024 (0.0408) | 0.250 (0.4101)
  Eosinophils, Day 7 | -0.039 (0.0498) | 0.325 (0.5869)
  Eosinophils, Day 10 | -0.009 (0.0628) | -0.055 (0.1485)
  Lymphocytes, Day 3 | 0.197 (0.2870) | -0.500 (0.3111)
  Lymphocytes, Day 7 | 0.190 (0.2514) | -0.525 (0.1485)
  Lymphocytes, Day 10 | 0.229 (0.2738) | -0.720 (0.5515)
  Monocytes, Day 3 | -0.030 (0.0876) | 0.170 (0.2121)
  Monocytes, Day 7 | -0.039 (0.1126) | 0.035 (0.1626)
  Monocytes, Day 10 | 0.056 (0.0774) | -0.005 (0.2192)
  Total Neutrophils, Day 3 | 0.181 (0.6097) | -0.080 (0.1273)
  Total Neutrophils, Day 7 | -0.003 (0.6304) | -0.155 (0.2192)
  Total Neutrophils, Day 10 | 0.831 (1.6043) | 0.405 (1.1384)
  White blood cell count, Day 3 | 0.34 (0.282) | -0.15 (1.061)
  White blood cell count, Day 7 | 0.11 (0.782) | -0.30 (1.131)
  White blood cell count, Day 10 | 1.11 (1.508) | -0.35 (1.626)

12. Primary Outcome: Change From Baseline in Hematology Parameters: Hemoglobin
Description: Blood samples for assessment of hematology parameter of hemoglobin was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: Safety population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Grams per deciliter
  Day 3 | 0.13 (0.637) | -0.30 (0.424)
  Day 7 | 0.06 (0.519) | 0.00 (0.424)
  Day 10 | -0.17 (0.446) | -0.15 (0.354)

13. Primary Outcome: Change From Baseline in Hematology Parameters: Mean Corpuscle Hemoglobin
Description: Blood samples for assessment of hematology parameter of mean corpuscle hemoglobin was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: Safety population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Picogram
  Day 3 | -0.03 (0.198) | 0.25 (0.495)
  Day 7 | 0.37 (0.411) | 0.30 (0.141)
  Day 10 | 0.00 (0.306) | 0.40 (0.424)

14. Primary Outcome: Change From Baseline in Hematology Parameters: Mean Corpuscle Volume
Description: Blood samples for assessment of hematology parameter of mean corpuscle volume was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: Safety Population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Femtoliter
  Day 3 | 1.0 (1.15) | 0.5 (0.71)
  Day 7 | 1.0 (1.63) | -0.5 (0.71)
  Day 10 | 1.7 (1.11) | 0.0 (1.41)

15. Primary Outcome: Change From Baseline in Hematology Parameters: Platelet Count
Description: Blood samples for assessment of hematology parameter of platelet count was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: Safety population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Cells per cubic millimeter
  Day 3 | 10428.6 (8847.92) | 5000.0 (21213.20)
  Day 7 | 15142.9 (29299.76) | 2500.0 (2121.32)
  Day 10 | 8000.0 (23860.71) | 9500.0 (37476.66)

16. Primary Outcome: Change From Baseline in Hematology Parameters: Red Blood Cell Count
Description: Blood samples for assessment of hematology parameter of red blood cell count was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: Safety Population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Million cells per microliter
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Million cells per microliter
  Day 3 | 0.03 (0.221) | -0.15 (0.071)
  Day 7 | -0.06 (0.151) | -0.05 (0.071)
  Day 10 | -0.09 (0.135) | -0.10 (0.141)

17. Primary Outcome: Change From Baseline in Hematology Parameters: Reticulocytes
Description: Blood samples for assessment of hematology parameter of reticulocytes was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: Safety Population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Giga cells per liter
  Day 3 | 5.51 (9.971) | 9.45 (1.768)
  Day 7 | 13.79 (27.361) | -6.50 (0.849)
  Day 10 | 13.79 (16.419) | 21.30 (35.497)

18. Primary Outcome: Change From Baseline in Clinical Chemistry Data: Albumin, Total Protein
Description: Blood samples for assessment of clinical chemistry parameters of albumin and total protein was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: Safety Population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Groups:
- GSK1265744 5 mg: Eligible participants received double-blind 5 mg GSK1265744 oral tablet once daily for 10 days.
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Grams per deciliter
  Albumin, Day 3 | 0.16 (0.162) | 0.00 (0.000)
  Albumin, Day 7: number analyzed (Participants) | 6 | 2
  Albumin, Day 7 | 0.08 (0.117) | 0.05 (0.071)
  Albumin, Day 10 | 0.06 (0.098) | 0.15 (0.071)
  Total protein, Day 3 | 0.24 (0.447) | 0.05 (0.212)
  Total protein, Day 7: number analyzed (Participants) | 6 | 2
  Total protein, Day 7 | 0.03 (0.294) | 0.10 (0.424)
  Total protein, Day 10 | -0.10 (0.342) | 0.10 (0.000)

19. Primary Outcome: Change From Baseline in Clinical Chemistry Data: Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatine Kinase, Lipase
Description: Blood samples for assessment of clinical chemistry parameters of alkaline phosphatase, alanine amino transferase, aspartate amino transferase, creatine kinase and lipase was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: Safety Population. Only those participants available at the indicated time points were analyzed. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Units per liter
Groups:
- GSK1265744 5 mg: Eligible participants received double-blind GSK1265744 5 mg tablet once daily for 10 days.
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Units per liter
  Alkaline phosphatase, Day 3 | 1.6 (3.10) | -3.5 (4.95)
  Alkaline phosphatase, Day 7: number analyzed (Participants) | 6 | 2
  Alkaline phosphatase, Day 7 | 0.5 (3.89) | -5.0 (0.00)
  Alkaline phosphatase, Day 10 | -2.4 (6.55) | -4.0 (2.83)
  Alanine amino transferase, Day 3 | 2.9 (6.41) | -4.0 (2.83)
  Alanine amino transferase, Day 7: number analyzed (Participants) | 6 | 2
  Alanine amino transferase, Day 7 | -0.2 (4.02) | -1.5 (9.19)
  Alanine amino transferase, Day 10 | 2.0 (4.12) | -2.5 (7.78)
  Aspartate amino transferase, Day 3 | -1.0 (4.28) | -2.0 (8.49)
  Aspartate amino transferase, Day 7: number analyzed (Participants) | 6 | 2
  Aspartate amino transferase, Day 7 | -1.0 (3.52) | -3.5 (7.78)
  Aspartate amino transferase, Day 10 | 0.4 (5.32) | -2.0 (5.66)
  Creatine kinase, Day 3 | -0.1 (11.42) | -29.5 (10.61)
  Creatine kinase, Day 7: number analyzed (Participants) | 6 | 2
  Creatine kinase, Day 7 | 27.7 (77.11) | -48.0 (42.43)
  Creatine kinase, Day 10 | 20.6 (42.97) | -40.5 (43.13)
  Lipase, Day 3 | 0.9 (8.91) | 4.0 (2.83)
  Lipase, Day 7 | -0.9 (17.22) | -1.0 (8.49)
  Lipase, Day 10 | 0.3 (14.42) | -2.0 (2.83)

20. Primary Outcome: Change From Baseline in Direct Bilirubin, Total Bilirubin, Calcium, Cholesterol, Creatinine, Glucose, High Density Lipoprotein (HDL) Cholesterol Direct, Low Density Lipoprotein (LDL) Cholesterol Calculation, Triglycerides, Urea/Blood Urea Nitrogen
Description: Blood samples for assessment of clinical chemistry parameters of direct bilirubin, total bilirubin, calcium, cholesterol, creatinine, glucose, HDL cholesterol direct, LDL cholesterol calculation, triglycerides,Urea/BUN was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Milligrams per deciliter
  Direct bilirubin, Day 3 | -0.04 (0.113) | -0.05 (0.071)
  Direct bilirubin, Day 7: number analyzed (Participants) | 6 | 2
  Direct bilirubin, Day 7 | -0.10 (0.126) | -0.05 (0.071)
  Direct bilirubin, Day 10 | -0.06 (0.053) | 0.00 (0.000)
  Total bilirubin, Day 3 | -0.06 (0.207) | -0.25 (0.354)
  Total bilirubin, Day 7: number analyzed (Participants) | 6 | 2
  Total bilirubin, Day 7 | -0.03 (0.186) | -0.40 (0.566)
  Total bilirubin, Day 10 | 0.00 (0.216) | -0.10 (0.141)
  Calcium, Day 3 | 0.13 (0.198) | 0.00 (0.141)
  Calcium, Day 7: number analyzed (Participants) | 6 | 2
  Calcium, Day 7 | 0.17 (0.207) | 0.05 (0.495)
  Calcium, Day 10 | -0.09 (0.254) | 0.20 (0.000)
  Cholesterol, Day 3 | 5.7 (8.90) | -7.5 (9.19)
  Cholesterol, Day 7: number analyzed (Participants) | 6 | 2
  Cholesterol, Day 7 | 16.2 (32.60) | 0.0 (1.41)
  Cholesterol, Day 10 | 4.0 (13.17) | 1.0 (2.83)
  Creatinine, Day 3 | 0.03 (0.049) | 0.05 (0.071)
  Creatinine, Day 7: number analyzed (Participants) | 6 | 2
  Creatinine, Day 7 | 0.05 (0.105) | 0.05 (0.071)
  Creatinine, Day 10 | 0.03 (0.076) | 0.05 (0.071)
  Glucose, Day 3 | 16.1 (28.35) | 2.0 (1.41)
  Glucose, Day 7: number analyzed (Participants) | 6 | 2
  Glucose, Day 7 | -16.5 (45.62) | 4.5 (3.54)
  Glucose, Day 10 | 0.1 (5.81) | -4.0 (0.00)
  HDL cholesterol, direct, Day 3 | -0.6 (2.44) | -1.5 (2.12)
  HDL cholesterol, direct, Day 7: number analyzed (Participants) | 6 | 2
  HDL cholesterol, direct, Day 7 | -0.2 (9.62) | 0.5 (0.71)
  HDL cholesterol, direct, Day 10 | 1.9 (4.56) | -2.0 (1.41)
  LDL cholesterol calculation, Day 3 | 6.7 (9.21) | -7.0 (12.73)
  LDL cholesterol calculation, Day 7: number analyzed (Participants) | 5 | 2
  LDL cholesterol calculation, Day 7 | -0.2 (9.93) | 3.5 (6.36)
  LDL cholesterol calculation, Day 10 | 1.6 (10.42) | -2.5 (16.26)
  Triglycerides, Day 3 | -1.9 (49.69) | 5.0 (4.24)
  Triglycerides, Day 7: number analyzed (Participants) | 6 | 2
  Triglycerides, Day 7 | 258.3 (636.46) | -20.5 (21.92)
  Triglycerides, Day 10 | 3.6 (39.59) | 28.5 (72.83)
  Urea/BUN, Day 3 | 1.4 (2.15) | -1.0 (5.66)
  Urea/BUN, Day 7: number analyzed (Participants) | 6 | 2
  Urea/BUN, Day 7 | 1.3 (3.27) | -2.5 (4.95)
  Urea/BUN, Day 10 | 0.7 (2.81) | -2.0 (0.00)

21. Primary Outcome: Change From Baseline in Clinical Chemistry Data: Chloride, Carbon Dioxide Content/Bicarbonate, Magnesium, Sodium, Potassium
Description: Blood samples for assessment of clinical chemistry parameters of chloride, carbon dioxide content/bicarbonate, magnesium, sodium and potassium was collected at Baseline, Day 3, 7 and 10. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 3, 7, 10
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Milliequivalents per liter
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Milliequivalents per liter
  Chloride, Day 3 | 0.0 (0.82) | 2.0 (0.00)
  Chloride, Day 7: number analyzed (Participants) | 6 | 2
  Chloride, Day 7 | -0.2 (2.79) | 2.0 (0.00)
  Chloride, Day 10 | -0.7 (2.69) | 2.0 (4.24)
  Carbon dioxide content/Bicarbonate, Day 3 | -0.9 (2.41) | -1.0 (0.00)
  Carbon dioxide content/Bicarbonate, Day 7: number analyzed (Participants) | 6 | 2
  Carbon dioxide content/Bicarbonate, Day 7 | -1.3 (1.63) | -2.0 (2.83)
  Carbon dioxide content/Bicarbonate, Day 10 | 0.6 (2.76) | -2.0 (2.83)
  Potassium, Day 3 | 0.20 (0.200) | 0.30 (0.141)
  Potassium, Day 7: number analyzed (Participants) | 6 | 2
  Potassium, Day 7 | 0.00 (0.245) | 0.20 (0.283)
  Potassium, Day 10 | 0.07 (0.368) | 0.05 (0.212)
  Magnesium, Day 3 | -0.04 (0.098) | 0.10 (0.000)
  Magnesium, Day 7: number analyzed (Participants) | 6 | 2
  Magnesium, Day 7 | -0.00 (0.089) | 0.10 (0.141)
  Magnesium, Day 10 | -0.04 (0.098) | 0.00 (0.141)
  Sodium, Day 3 | -0.4 (1.62) | 0.5 (0.71)
  Sodium, Day 7: number analyzed (Participants) | 6 | 2
  Sodium, Day 7 | 0.3 (2.50) | 0.5 (0.71)
  Sodium, Day 10 | -0.4 (1.62) | 0.5 (2.12)

22. Primary Outcome: Number of Participants With Urinalysis Data
Description: Samples for urinalysis assessment was collected on Day 1, Day 3 and Day 10. Urinalysis parameters included urine bilirubin, urine occult blood, urine glucose, urine ketones, urine nitrite, urine pH, urine protein, urine specific gravity and urine leukocyte esterase test for detecting white blood cell.
Time Frame: Day 1 to Day 10
Population: Safety Population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Participants
  Day 1, Urine Bilirubin, Negative | 7 | 2
  Day 1, Urine Occult Blood, Negative | 7 | 2
  Day 1, Urine Glucose, Negative | 7 | 2
  Day 1, Urine Ketones, Negative | 7 | 2
  Day 1, Urine Nitrite, Negative | 6 | 2
  Day 1, Urine Nitrite, Positive | 1 | 0
  Day 1, Urine pH, 5.5 | 2 | 1
  Day 1, Urine pH, 6 | 4 | 1
  Day 1, Urine pH, 6.5 | 1 | 0
  Day 1, Urine Protein, Negative | 7 | 2
  Day 1, Urine Specific Gravity, 1.006 | 1 | 0
  Day 1, Urine Specific Gravity, 1.014 | 0 | 1
  Day 1, Urine Specific Gravity, 1.015 | 0 | 1
  Day 1, Urine Specific Gravity, 1.017 | 1 | 0
  Day 1, Urine Specific Gravity, 1.019 | 2 | 0
  Day 1, Urine Specific Gravity, 1.021 | 1 | 0
  Day 1, Urine Specific Gravity, 1.025 | 1 | 0
  Day 1, Urine Specific Gravity, 1.03 | 1 | 0
  Day 1, ULET for white blood cell, Negative | 7 | 2
  Day 3, Urine Bilirubin, Negative | 7 | 2
  Day 3, Urine Occult Blood, Negative | 6 | 2
  Day 3, Urine Occult Blood, 1+ | 1 | 0
  Day 3, Urine Glucose, 3+ | 1 | 0
  Day 3, Urine Glucose, Negative | 6 | 2
  Day 3, Urine Ketones, Negative | 7 | 2
  Day 3, Urine Nitrite, Negative | 6 | 2
  Day 3, Urine Nitrite, Positive | 1 | 0
  Day 3, Urine pH, 5.5 | 4 | 1
  Day 3, Urine pH, 6 | 2 | 1
  Day 3, Urine pH, 6.5 | 1 | 0
  Day 3, Urine Protein, Negative | 6 | 2
  Day 3, Urine Protein, Trace | 1 | 0
  Day 3, Urine Specific Gravity, 1.016 | 1 | 0
  Day 3, Urine Specific Gravity, 1.017 | 1 | 1
  Day 3, Urine Specific Gravity, 1.018 | 0 | 1
  Day 3, Urine Specific Gravity, 1.021 | 2 | 0
  Day 3, Urine Specific Gravity, 1.022 | 1 | 0
  Day 3, Urine Specific Gravity, 1.027 | 1 | 0
  Day 3, Urine Specific Gravity, 1.03 | 1 | 0
  Day 3, ULET for white blood cell, 2+ | 1 | 0
  Day 3, ULET for white blood cell, Negative | 6 | 2
  Day 10, Urine Bilirubin, Negative | 7 | 2
  Day 10, Urine Occult Blood, 2+ | 1 | 0
  Day 10, Urine Occult Blood, Negative | 6 | 2
  Day 10, Urine Glucose, Negative | 7 | 2
  Day 10, Urine Ketones, Negative | 7 | 2
  Day 10, Urine Nitrite, Negative | 6 | 2
  Day 10, Urine Nitrite, Positive | 1 | 0
  Day 10, Urine pH, 5.5 | 0 | 1
  Day 10, Urine pH, 6 | 4 | 1
  Day 10, Urine pH, 6.5 | 3 | 0
  Day 10, Urine Protein, Negative | 5 | 2
  Day 10, Urine Protein, Trace | 2 | 0
  Day 10, Urine Specific Gravity, 1.009 | 0 | 1
  Day 10, Urine Specific Gravity, 1.016 | 0 | 1
  Day 10, Urine Specific Gravity, 1.02 | 1 | 0
  Day 10, Urine Specific Gravity, 1.021 | 1 | 0
  Day 10, Urine Specific Gravity, 1.023 | 1 | 0
  Day 10, Urine Specific Gravity, 1.025 | 2 | 0
  Day 10, Urine Specific Gravity, 1.027 | 1 | 0
  Day 10, Urine Specific Gravity, 1.03 | 1 | 0
  Day 10, ULET for white blood cell, Negative | 7 | 2

23. Primary Outcome: Change From Baseline in Vital Sign: Systolic and Diastolic Blood Pressure
Description: Systolic and diastolic blood pressure was measured at Baseline (Day 1 pre-dose), 2 hour post dose on Day 1, pre-dose on Day 4, 7, 10 and 2 hours post dose on Day 10. Baseline was defined at Day 1 pre-dose. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1, pre-dose) and Day 1 (2 hours post dose), 4, 7, 10
Population: Safety population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Millimeters of mercury (mmHg)
  Systolic blood pressure, Day 1, 2 Hours | 1.2 (8.59) | 5.8 (0.35)
  Systolic blood pressure, Day 4, Pre dose | 1.8 (9.16) | 5.8 (3.18)
  Systolic blood pressure, Day 7, Pre dose | -2.5 (11.22) | -4.3 (8.84)
  Systolic blood pressure, Day 10, Pre dose | 0.6 (19.19) | 19.8 (14.50)
  Systolic blood pressure, Day 10, 2 Hours | -0.2 (10.59) | 13.3 (4.60)
  Diastolic blood pressure, Day 1, 2 Hours | -5.7 (5.76) | -0.5 (2.12)
  Diastolic blood pressure, Day 4, Pre dose | -2.4 (8.91) | -2.5 (10.61)
  Diastolic blood pressure, Day 7, Pre dose | -1.6 (9.28) | -5.0 (15.56)
  Diastolic blood pressure, Day 10, Pre dose | -5.4 (13.85) | 8.5 (14.85)
  Diastolic blood pressure, Day 10, 2 Hours | -2.4 (6.82) | 6.5 (9.19)

24. Primary Outcome: Change From Baseline in Vital Sign: Heart Rate
Description: Heart rate was measured at Baseline (Day 1 pre-dose), 2 hour post dose on Day 1, pre-dose on Day 4, 7, 10 and 2 hours post dose on Day 10. Baseline was defined at Day 1 pre-dose. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1, pre-dose) and Day 1 (2 hours post dose), 4, 7, 10
Population: Safety population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Beats per minute
  Day 1, 2 Hours | -7.0 (2.10) | -5.8 (4.60)
  Day 4, Pre dose | 5.3 (6.24) | -5.8 (1.06)
  Day 7, Pre dose | 6.3 (5.71) | -1.8 (1.77)
  Day 10, Pre dose | 0.0 (6.74) | 5.8 (4.60)
  Day 10, 2 Hours | -7.6 (5.12) | -10.8 (3.18)

25. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters
Description: All ECGs were obtained after a minimum 10 minute rest in a semi-supine position. The 12-lead ECGs were obtained at Baseline (Day 1 pre-dose), 2 hour post dose on Day 1, pre-dose on Day 4, 7, 10 and 2 hours post dose on Day 10 using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and Bazett's correction (QTcB) and Fridericia correction (QTcF) intervals. Baseline was defined at Day 1 pre-dose. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1, pre-dose) and Day 1 (2 hours post dose), 4, 7, 10
Population: Safety population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Milliseconds (msec)
  PR, Day 1, 2 Hours | 0.0 (1.83) | 1.0 (2.83)
  PR, Day 4, Pre dose | 4.0 (5.42) | 5.0 (11.31)
  PR, Day 7, Pre dose | -0.9 (4.67) | 0.0 (12.73)
  PR, Day 10, Pre dose | -1.7 (3.04) | 0.0 (9.90)
  PR, Day 10, 2 Hours | 4.3 (10.09) | 4.0 (12.73)
  QRS, Day 1, 2 Hours | -0.7 (3.68) | 1.5 (0.71)
  QRS, Day 4, Pre dose | 0.7 (2.36) | -3.5 (12.02)
  QRS, Day 7, Pre dose | -0.1 (4.26) | 3.5 (2.12)
  QRS, Day 10, Pre dose | 1.0 (5.07) | 0.5 (3.54)
  QRS, Day 10, 2 Hours | -0.7 (8.99) | 5.5 (4.95)
  QT, Day 1, 2 Hours | 18.1 (8.07) | 27.0 (24.04)
  QT, Day 4, Pre dose | -10.7 (20.93) | 5.0 (7.07)
  QT, Day 7, Pre dose | -13.6 (13.13) | 11.0 (1.41)
  QT, Day 10, Pre dose | -3.3 (14.14) | -11.0 (24.04)
  QT, Day 10, 2 Hours | 19.0 (22.15) | 25.0 (24.04)
  QTcB, Day 1, 2 Hours | 0.2 (13.50) | 6.0 (4.09)
  QTcB, Day 4, Pre dose | 2.0 (16.15) | -17.9 (2.20)
  QTcB, Day 7, Pre dose | -0.0 (16.95) | -9.0 (25.73)
  QTcB, Day 10, Pre dose | 1.4 (16.59) | -15.6 (10.35)
  QTcB, Day 10, 2 Hours | -2.4 (12.35) | -18.1 (0.42)
  QTcF, Day 1, 2 Hours | 6.4 (11.45) | 13.3 (11.06)
  QTcF, Day 4, Pre dose | -2.4 (14.27) | -10.0 (4.05)
  QTcF, Day 7, Pre dose | -4.7 (13.05) | -2.0 (16.30)
  QTcF, Day 10, Pre dose | -0.2 (13.17) | -13.9 (15.19)
  QTcF, Day 10, 2 Hours | 4.9 (13.62) | -3.4 (7.99)

26. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA
Description: Plasma for quantitative HIV-1 RNA was collected on Day 1, 2, 3, 4, 7, 8, 9, 10 and 11. On Days 1, 10 and 11, two samples for HIV-1 RNA were collected between 5-20 minutes apart to reduce sample variability. An HIV-1 RNA PCR assay with a LLOD of 50 copies/mL (ultrasensitive assay) was used for post-baseline assessments. An HIV-1 RNA PCR assay with a LLOD of 400 copies/mL (standard assay) was used for screening and Baseline assessments and included a re-test with and ultrasensitive assay for all Baseline values below the LLOD. Baseline was defined at Day 1 (pre-dose). The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1 pre-dose) and Day 1 (post dose), 2, 3, 4, 7, 8, 9, 10
Population: ITT population. Only those participants available at the indicated time points were analyzed. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Log10 copies/mL
  Day 1: number analyzed (Participants) | 7 | 1
  Day 1 | 0.000 (0.0000) | 0.000 (NA) — Only one participant was analyzed.
  Day 2 | -0.126 (0.2255) | 0.058 (0.2303)
  Day 3 | -0.618 (0.1341) | -0.299 (0.2737)
  Day 4 | -0.830 (0.2424) | -0.146 (0.0580)
  Day 7 | -1.577 (0.5498) | -0.168 (0.1264)
  Day 8 | -1.935 (0.4717) | -0.146 (0.2779)
  Day 9 | -2.013 (0.4192) | -0.007 (0.1960)
  Day 10 | -2.160 (0.2810) | -0.158 (0.1930)

27. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA to Nadir Over 11 Days
Description: Plasma for quantitative HIV-1 RNA was collected on Day 1, 2, 3, 4, 7, 8, 9, 10 and 11. On Days 1, 10 and 11, two samples for HIV-1 RNA was collected between 5-20 minutes apart to reduce sample variability. An HIV-1 RNA PCR assay with a LLOD of 50 copies/mL (ultrasensitive assay) was used for post-baseline assessments. An HIV-1 RNA PCR assay with a LLOD of 400 copies/mL (standard assay) was used for screening and Baseline assessments and included a re-test with and ultrasensitive assay for all Baseline values below the LLOD. Nadir was the maximum change from Baseline in plasma HIV-1 RNA. Baseline was defined at Day 1 (pre-dose). The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 11
Population: ITT population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
log10 copies/mL | -2.199 (0.2491) | -0.418 (0.1058)
Statistical Analysis 1: Comparison: GSK1265744 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA with treatment as fixed effect, and baseline HIV-1 RNA as covariate; Mean Difference (Net) = -1.804, 95% CI 2-sided [-2.173 to -1.436]

28. Secondary Outcome: Plasma HIV-1 RNA Rate of Decline (Slope) Over 11 Days
Description: Plasma for quantitative HIV-1 RNA was collected on Day 1, 2, 3, 4, 7, 8, 9, 10 and 11. On Days 1, 10 and 11, two samples for HIV-1 RNA was collected between 5-20 minutes apart to reduce sample variability. An HIV-1 RNA PCR assay with a LLOD of 50 copies/mL (ultrasensitive assay) was used for post-baseline assessments. An HIV-1 RNA PCR assay with a LLOD of 400 copies/mL (standard assay) was used for screening and Baseline assessments and included a re-test with and ultrasensitive assay for all Baseline values below the LLOD. Estimated mean rate of decline (i.e., slope of day) with corresponding 90% confidence interval was provided for each treatment.
Time Frame: Up to Day 10
Population: ITT population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (90% Confidence Interval); unit: log10 copies per mL per day
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
log10 copies per mL per day | -0.2313 [-0.2513 to -0.2113] | 0.0013 [-0.0233 to 0.0259]
Statistical Analysis 1: Comparison: GSK1265744 5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

29. Secondary Outcome: Number of Participants With HIV-1 RNA<400 Copies/mL
Description: Plasma for quantitative HIV-1 RNA was collected on Day 1, 2, 3, 4, 7, 8, 9, 10 and 11. On Days 1, 10 and 11, two samples for HIV-1 RNA was collected between 5-20 minutes apart to reduce sample variability. An HIV-1 RNA PCR assay with a LLOD of 50 copies/mL (ultrasensitive assay) was used for post-baseline assessments. An HIV-1 RNA PCR assay with a LLOD of 400 copies/mL (standard assay) was used for screening and Baseline assessments and included a re-test with and ultrasensitive assay for all Baseline values below the LLOD. assessments and included a re-test with and ultrasensitive assay for all Baseline values below the LLOD. Only categories with data available at the indicated time points have been presented. Categories with null values for all the arms have not been presented.
Time Frame: Up to Day 11
Population: ITT population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Participants
  Day 7 | 2 | 0
  Day 8 | 4 | 0
  Day 9 | 4 | 0
  Day 10 | 5 | 0
  Day 11 | 5 | 0

30. Secondary Outcome: Number of Participants With HIV-1 RNA<50 Copies/mL
Description: as for outcome 29
Time Frame: Up to Day 11
Population: ITT population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Participants
  Day 8 | 2 | 0
  Day 9 | 3 | 0
  Day 10 | 2 | 0
  Day 11 | 2 | 0

31. Secondary Outcome: Change From Baseline in CD4+ Cell Count to Day 11
Description: Whole venous blood samples was obtained from each participant for the analysis of lymphocyte subsets by flow cytometry on Day 1 and Day 11. Baseline was defined at Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) and Day 11
Population: ITT population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | GSK1265744 5 mg | Placebo
Number analyzed (Participants) | 7 | 2
Cells per cubic millimeter | 71.0 (56.62) | -84.0 (145.66)

32. Secondary Outcome: Pre-morning Dose Concentrations (C0) on Day 2 Through 10 to Assess the Achievement of Steady State of GSK1265744 Following Repeat Administration
Description: Steady state is said to be reached, when the pre-dose concentration slope estimate is close to zero. The data for pre-dose concentration on Day 1 24 hours (Day 2) through Day 10 has been presented.
Time Frame: Day 1 24 hours (Day 2), Pre-dose on Days 3, 4, 7, 8, 9 and 10
Population: ITT population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 7
µg/mL
  DAY 1, 24 hours (Day 2) | 0.2363 (0.06884)
  DAY 3, Pre-dose | 0.3539 (0.12999)
  DAY 4, Pre-dose | 0.4128 (0.15566)
  DAY 7, Pre-dose | 0.5239 (0.11899)
  DAY 8, Pre-dose | 0.5744 (0.17622)
  DAY 9, Pre-dose | 0.5688 (0.16880)
  DAY 10, Pre-dose | 0.5654 (0.20609)

33. Secondary Outcome: Accumulation Ratios for AUC, Cmax, and Ctau
Description: The accumulation ratio was calculated as the ratio of AUC(0-τ), Cmax, and Ctau on Day 10 to AUC(0-24), Cmax, and C24 on Day 1 for each participant. The ratio of geometric least square means of each parameter on Day 10 to Day 1 was presented along with 90% confidence interval.
Time Frame: Days 1 and 10
Population: PK/ Pharmacodynamic (PD) Summary Population included participants who met the criteria for both ITT Population and PK Summary Population. GSK1265744 30 mg arm is from study ITZ111451 that was used only for dose proportionality assessments.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | GSK1265744 5 mg
Number analyzed (Participants) | 7
Ratio
  Accumulation Ratio AUC | 2.355 [2.086 to 2.658]
  Accumulation Ratio Cmax | 1.961 [1.684 to 2.283]
  Accumulation Ratio Ctau | 2.483 [2.141 to 2.880]

34. Secondary Outcome: Day 1 AUC(0-24) at Different Doses for the Assessment of Dose Proportionality Using Power Model
Description: Data from GSK1265744 30 mg in HIV participants (Study ITZ111451 part C HIV cohort, NCT00659191) was combined with data from this study to access dose proportionality. Dose proportionality of GSK1265744 PK parameters was assessed following single dose administration on Day 1 (AUC[0-24]) using the power model. The mean slope and corresponding 90% confidence interval has been presented.
Time Frame: Day 1
Population: PK Summary Population.
Measure: Mean (90% Confidence Interval); unit: hr*µg/mL/mg
Groups:
- Pooled GSK1265744: Eligible participants received double-blind GSK1265744 5 mg oral tablet once daily for 10 days in the current study ITZ112929 and repeat doses of GSK1265744 30 mg (6x5 mg) oral tablets once daily for 10 days in study ITZ111451.
Arm/Group | Pooled GSK1265744
Number analyzed (Participants) | 15
hr*µg/mL/mg | 0.952 [0.802 to 1.101]

35. Secondary Outcome: Day 1 Cmax and C24 at Different Doses for the Assessment of Dose Proportionality Using Power Model
Description: Data from GSK1265744 30 mg in HIV participants (Study ITZ111451 part C HIV cohort, NCT00659191) was combined with data from this study to access dose proportionality. Dose proportionality of GSK1265744 PK parameters was assessed following single dose administration on Day 1 (Cmax, and C24) using the power model. The mean slope and corresponding 90% confidence interval has been presented.
Time Frame: Day 1
Population: PK Summary Population.
Measure: Mean (90% Confidence Interval); unit: μg/mL/mg
Arm/Group | Pooled GSK1265744
Number analyzed (Participants) | 15
μg/mL/mg
  Cmax | 0.950 [0.812 to 1.088]
  C24 | 0.949 [0.777 to 1.121]

36. Secondary Outcome: Day 10 AUC(0-tau) at Different Doses for the Assessment of Dose Proportionality Using Power Model
Description: Data from GSK1265744 30 mg in HIV participants (Study ITZ111451 part C HIV cohort, NCT00659191) was combined with data from this study to access dose proportionality. Dose proportionality of GSK1265744 PK parameters was assessed following a repeat dose administration on Day 10 (AUC[0-tau]) using the power model. The mean slope and corresponding 90% confidence interval has been presented.
Time Frame: Day 10
Population: PK Summary Population.
Measure: Mean (90% Confidence Interval); unit: hr*µg/mL/mg
Arm/Group | Pooled GSK1265744
Number analyzed (Participants) | 15
hr*µg/mL/mg | 0.988 [0.841 to 1.135]

37. Secondary Outcome: Day 10 Cmax, C0 and Ctau at Different Doses for the Assessment of Dose Proportionality Using Power Model
Description: Data from GSK1265744 30 mg in HIV participants (Study ITZ111451 part C HIV cohort, NCT00659191) was combined with data from this study to access dose proportionality. Dose proportionality of GSK1265744 PK parameters was assessed following a repeat dose administration on Day 10 (Cmax, Ctau and C0) using the power model. The mean slope and corresponding 90% confidence interval has been presented.
Time Frame: Day 10
Population: PK Summary Population.
Measure: Mean (90% Confidence Interval); unit: µg/mL/mg
Arm/Group | Pooled GSK1265744
Number analyzed (Participants) | 15
µg/mL/mg
  Cmax | 1.025 [0.903 to 1.147]
  C0 | 0.936 [0.761 to 1.110]
  Ctau | 0.980 [0.808 to 1.151]

ADVERSE EVENTS:
Time Frame: Up to follow-up visit (Day 25±1)
Description: Safety Population was used.
Groups:
- Placebo: Eligible participants received double-blind Placebo matching 5 mg GSK1265744 oral tablet once daily for 10 days.
Arm/Group | GSK1265744 30 mg | GSK1265744 5 mg | Placebo | Optimized Therapy
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/2 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 0/7 | 2/2 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1265744 30 mg (N=8) | GSK1265744 5 mg (N=7) | Placebo (N=2) | Optimized Therapy (N=8)
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.